

# **Appendix A: Study Protocol**

# Transitioning Youth Out of Homelessness 2.5: A Co-Designed Strengths-Based Leadership Program for Young People Transitioning Out of Homelessness

#### **Abstract**

**Background**: This project builds on our current community-based randomized clinical trial (Transitioning Youth Out of Homelessness 2.0) utilizing coaching and a co-designed leadership guide to target identity capital (purpose, control, self-efficacy, and self-esteem) for youth transitioning out of homelessness (all participants are also receiving rent subsidies). Based on preliminary feedback from study youth and coaches involved in the intervention arm, we plan to modify the leadership guide and pilot it in the form of an in-person, four-week leadership program (vs. independent learning in our current study).

**Objectives:** The overarching objective of this mixed methods pilot project is to co-develop and test a strengths-based leadership program targeting identity capital for youth (16 - 24 years of age) transitioning out of homelessness. Specifically, the objectives are to:

- 1. Modify the leadership guide being used in our current study so it can be delivered as an in-person leadership program.
- **2.** Co-develop and pilot a four-week, strengths-based leadership program for young people transitioning out of homelessness.
- **3.** Determine the feasibility and acceptability of the leadership guide when delivered as a four-week, in-person program (as opposed to independent learning in our current study).
- **4.** Examine whether self-reported measures of identity capital and knowledge of program material show improvement immediately post-program compared to baseline.
- **5.** Explore whether there are differences in outcomes by sub-groups (e.g., gender, age, identification as 2SLGBTQ+, child welfare involvement) and/or program participation levels.

**Methods:** This study will employ a mixed method design embedded within a Community Based Participatory Action Research framework. *Phase One (Objectives 1 & 2):* An established team of

two coaches and four youth lived expert advisors will collaborate with a Toronto-based high school teacher on modifying the guide and co-developing the leadership program. *Phase Two (Objective 2):* Participants (n = 30) will be recruited from our community partner agencies. Two four-week leadership programs (15 youth per program) will be led by coaches from our current study with our youth advisors participating as paid leadership interns. Data collection will occur at baseline (baseline demographic questionnaire; identity capital questionnaire; knowledge assessment questionnaire) and immediately post-program (identity capital questionnaire; knowledge assessment questionnaire; program feedback questionnaire; focus group). We will also track program session attendance. *Phase Three (Objectives 3, 4 & 5):* Quantitative questionnaires and program attendance will be examined using descriptive statistics and non-parametric or t-tests and Cohen's d effect size. Qualitative focus groups (primarily centred around acceptability) will be explored using reflexive thematic analysis with a critical social theoretical lens.

**Significance:** If this modified delivery of the leadership guide shows promise, we plan to incorporate it into a national scale-up alongside rent subsidies and coaching.

# 1. Background and Rationale

Drivers into youth homelessness are well documented and include multiple adverse childhood experiences, poverty, discrimination, and child welfare involvement (Abramovich, 2016; Centrepoint, 2022; Crandall et al., 2019; Dej, 2020; Gaetz et al., 2016; Karabanow, 2004; Karabanow et al., 2016; Liu et al., 2021; Morton et al., 2018; Samuels et al., 2019). The impact of being failed by people and systems intended to nurture and support have profound impacts on the health and well-being of these inequitably served youth (Abramovich, 2016; Bonakdar et al., 2023; Brueckner et al., 2011; Crandall et al., 2019; Dej, 2020; Gaetz et al., 2016; Karabanow et al., 2016; Kidd et al., 2016; Kidd et al., 2021; Kozloff et al., 2016; Liu et al., 2021; Mayock et al., 2011; Samuels et al., 2019; Thulien et al., 2018). For example, a 2019 pan-Canadian survey of 1,375 young people accessing supports within the youth homelessness system (e.g., shelter drop-in services) reported 74% of youth were experiencing high degrees of mental health distress (e.g., anxiety and/or depression) and 35% had tried to commit suicide at least once (Kidd et al., 2021). Levels of mental health distress and suicidality were the highest among younger

respondents, those with an earlier age of first homelessness, and those who identified as a woman/girl, Indigenous, and/or two-spirit, lesbian, gay, bisexual, transgender, or queer (2SLGBTQ+; Kidd et al., 2021). A notable 61% reported involvement with child protective services, with just under half (48%) reporting that they did not receive any help regarding a suitable plan for where they could go or how they could support themselves after exiting the child welfare system (Bonakdar et al., 2023).

The problem of no suitable plan for long-term, equitable social and economic inclusion (i.e., supports beyond housing and welfare payments) is emerging as a critical societal issue for young people attempting to transition away from homelessness. Research from the small but growing body of longitudinal studies on post-homelessness experiences highlights that, despite the attainment of relative housing stability and irrespective of the type of housing acquired (market rent with limited or no social service supports vs. subsidized with social services supports), too many youth are surviving, not thriving – struggling with poverty-level incomes, feelings of purposelessness, loneliness, "outsiderness", meaninglessness, hopelessness, and a sense of being stuck (Brueckner et al., 2011; Karabanow et al., 2016; Kidd et al., 2016; Kozloff et al., 2016; Mayock et al., 2011; Thulien et al., 2018, p. 6). Moreover, there is an extremely limited evidence base regarding effective and rigorous interventions for this population (Morton et al., 2020), especially when it comes to inclusion health – an emergent approach that aims to address extreme health and social inequities (Luchenski et al., 2018).

This project builds on our 2.5-year community-based pilot mixed method randomized clinical trial of rent subsidies and mentorship for youth exiting homelessness (Transitioning Youth Out of Homelessness 1.0; Thulien et al., 2019). While we were unable to prove that youth receiving rent subsidies and mentorship had significantly better socioeconomic inclusion outcomes compared to the group who received rent subsidies only, there were signals from our quantitative and qualitative data that connecting with informal mentors – people outside the study who played "coach-like" roles (e.g., asking powerful, future-oriented questions vs. simply providing advice) – was key to fostering socioeconomic inclusion (proxy indicators of socioeconomic inclusion encompassed measures such as community integration, self-esteem, and engagement in education, employment, and training; Thulien et al., 2022; Thulien et al., 2023).

Drawing on 71 in-depth interviews conducted by Dr. Naomi Thulien over the 2.5-year study period, the study also highlighted the crucial role of identity capital – a sense of purpose, control, self-efficacy, and self-esteem – as an important mediator of socioeconomic inclusion (Thulien et al., 2023). When people with limited identity capital encounter challenges, they are more likely to give up and take the path of least resistance (Côté, 2016). For study participants, this inequitable fostering of identity capital meant living in the legacy of their past (e.g., a sense of powerlessness over their futures) and becoming trapped in the "fog" of exclusion (Thulien et al., 2023, p. 5).

Building on these findings, our team of youth with lived expertise, community partners, and researchers, developed Transitioning Youth Out of Homelessness (TYOH) 2.0 – a pilot mixed method randomized clinical trial of rent subsidies and coaching along with a co-designed leadership guide for youth exiting homelessness (ClinicalTrials.gov, 2023). Briefly, all participants (n = 40) receive rent subsidies and half are randomly assigned a solution-focused coach and a leadership guide which was co-designed with youth who have experienced homelessness (including several youth from the TYOH 1.0 study). Young people in the intervention group are expected to engage one-on-one with their coach, and independently with the leadership guide for one year. We are trying to understand if this more deliberate targeting of identity capital (alongside rent subsidies) will show promise as a way to improve socioeconomic inclusion outcomes. Our goal is to use these findings to conduct a larger national study.

Preliminary qualitative feedback from TYOH 2.0 coaches and study participants is that, while the co-designed leadership guide is a tremendous resource, it is hard for youth to independently engage with the material (e.g., showing up to one-on-one coaching sessions with minimal/no engagement with the leadership guide beforehand). We have also had enthusiastic feedback from teachers in the Ontario Education and Community Partnership Program (ECPP) – a program designed to reach youth not engaged in traditional school settings (e.g., shelter-based schools) – that the guide has tremendous potential for use in an ECPP setting (e.g., high school credits for guide completion). Given our plan to incorporate the leadership guide into a TYOH 2.0 national scale-up (alongside rent subsidies and coaching), we plan to collaborate with our established youth advisors on modifying the leadership guide and make it more engaging, align it with the

Ontario Ministry of Education core high school learning competencies, and pilot it in the form of an in-person, four-week leadership program with youth who are transitioning out of homelessness.

# 1.1. Objectives

The overarching objective of this mixed methods pilot project is to co-develop and test a strengths-based leadership program targeting identity capital for youth (16 - 24 years old) transitioning out of homelessness. Specifically, the objectives are to:

- 1. Modify the leadership guide currently being used in TYOH 2.0 so it can be delivered as an in-person leadership program.
- **2.** Co-develop and pilot a four-week, strengths-based leadership program for young people transitioning out of homelessness.
- **3.** Determine the feasibility and acceptability of the leadership guide when delivered as a four-week, in-person program (as opposed to independent learning in the TYOH 2.0 study).
- **4.** Examine whether self-reported measures of identity capital and knowledge of program material show improvement immediately post-program compared to baseline.
- **5.** Explore whether there are differences in outcomes by sub-groups (e.g., gender, age, identification as 2SLGBTQ+, child welfare involvement) and/or program participation levels.

## 2. Methodology and Methods

This study and the past five years of collaborative work in this area is grounded in a commitment to centring voices of youth with lived expertise as well as responding to priorities defined by community partners. The overall study draws on key principles of community-based participatory action research (CBPAR) and the qualitative component is framed with a critical social theoretical lens (Israel et al., 2018; Kirkham & Anderson, 2010; Moosa-Mitha, 2015; Strega, 2015):

• Research participants are viewed as experts in their own lives.

- Focus on highlighting how inequitable social structures of power including the intersection of factors such as race, class, and gender – play out in the lives of participants.
- Search for examples of resilience and agency despite socio-structural inequities.
- Concerted effort to acknowledge and reduce power imbalances between researchers and the community.
- Equal value placed on academic knowledge and experiential knowledge.
- Commitment to co-producing practical, actionable data to build community capacity and improve the lives of research participants.
- Duty to remain invested with the community beyond the life of the research project.

## 2.1. Trial Design

This pilot study will employ a mixed methods design embedded within a CBPAR framework. The study will be conducted collaboratively with three long-term community partners who serve youth who are experiencing or have experienced homelessness: 1) Covenant House Toronto (Toronto, ON); 2) The RAFT (St. Catharines, ON); and 3) StepStones for Youth (Toronto, ON). We will prospectively register this trial on Clinicaltrials.gov once we receive Unity Health Toronto Research Ethics Board approval.

# 2.2. Eligibility Criteria

Eligible young people aged 16 - 24 years who have transitioned out of homelessness (e.g., no longer living in a shelter or couch surfing), defined as 3 consecutive months within the past 12 months, will be identified by our community partners (note: for the purpose of this study, youth living in foster care will be considered homeless). This age mandate was chosen because this is the age group served by our community partners. We have chosen to target the first year of exiting homelessness because our collective experience has shown that this can be a particularly precarious time for youth in terms of mental health challenges and risk of (re)experiencing homelessness (even if youth have attempted exits in the past).

In addition to the above age and housing **inclusion** criteria, study participants must:

• Be able to provide free and informed consent.

- Be able to understand English (leadership program and data collection will be conducted in English).
- Have experienced homelessness (e.g., unstable housing arrangements including shelter stays, foster care, and couch surfing) for 3 consecutive months in the past 12 months.
- Be able to consistently attend the four-week leadership program.

Young people will be **excluded** from the study if they are:

• Enrolled in a program or study with similar features to the TYOH 2.5 leadership program.

#### 2.3. Intervention

An established TYOH 2.0 core team of two coaches and four youth lived expert advisors will collaborate with Dr. Thulien and the TYOH 2.5 research team on modifying the leadership guide currently being used in the TYOH 2.0 study (Appendix B: Leadership Guide) so it can be delivered as an in-person, four-week (two sessions/week) leadership program. They will be joined by a high school teacher (and former ECPP teacher at Covenant House Toronto) who will help align the guide with the Ontario Ministry of Education core high school learning competencies for potential consideration of high school credits for leadership program completion (note: we will unlikely be able to guarantee a high school credit at this pilot stage, but plan to develop the guide with this goal in mind for our planned scale-up).

At the same time the leadership guide is being modified, the team will collaborate on how best to deliver material during the four-week, in-person program (Table 1). The leadership sessions will be held in a public library, last approximately three hours, and be led by coaches from our current study with our youth advisors participating as paid leadership interns. Participants will be paid \$25.00/hour for attending the program and receive a certificate upon program completion.

Table 1. TYOH 2.5 Leadership Program\*

| SESSION | KEY FOCUS/ACTIVITES |
|---|---|
| 1 | Consent forms |
| (Week One) | Baseline questionnaires |
| | <ul> <li>Examine link between mindfulness and purpose</li> </ul> |
| 2 | Explore core values |
| (Week One) | • Create a vision board |
| 3 | Examine link between core values and mood |
| (Week Two) | • Create a daily routine |
| 4 | Discover strategies to develop good habits |
| (Week Two) | <ul> <li>Understand difference between excellence and perfection</li> </ul> |
| ONE WEEK BREAK | |
| 5 | Review pre-break key learnings |
| (Week Three) | <ul> <li>Explore link between identity and behaviour</li> </ul> |
| | • Develop strategies to live in alignment with positive identity |
| 6 | Examine growth mindset vs. fixed mindset |
| (Week Three) | <ul> <li>Explore link between purpose and connecting with others</li> </ul> |
| 7 | Explore concept of scarcity |
| (Week Four) | • Understand link between vulnerability, courage, and worthiness |
| 8 | Review and share key learnings |
| (Week Four) | <ul> <li>Discuss next steps</li> </ul> |
| | <ul> <li>Complete questionnaires</li> </ul> |
| | <ul> <li>Celebration meal</li> </ul> |
| | • Focus group |

<sup>\*</sup>Note: A more comprehensive/detailed session-by-session agenda will be developed in collaboration with youth advisors during the co-design stage.

# 2.4. Study Outcomes

The primary outcomes for this pilot program are feasibility and acceptability (Table 2). Secondary outcomes include knowledge of program material and identity capital (Table 2).

Exploratory outcomes are differences in primary/secondary outcomes by sub-groups (e.g., gender, age, identification as 2SLGBTQ+, child welfare involvement) and/or program participation levels (Table 2).

Table 2. TYOH 2.5 Key Outcome Variables and Instruments

| <b>Key Outcome Variables</b> | Instruments | Collection |
|---|---|---|
| | | Timepoints* |
| <b>Primary Outcomes</b> | | |
| Feasibility and | Recruitment and enrollment metrics | Т0 |
| Acceptability | Session attendance | T1/T2 |
| | Dropout metrics | T1/T2 |
| | Focus group | T2 |
| | Composite program feedback | T2 |
| | questionnaire | |
| <b>Secondary Outcomes</b> | | |
| Knowledge of Program | Composite knowledge assessment | T1/T2 |
| Material | scale | |
| Identity Capital | Multi-Measure Agentic Personal | T1/T2 |
| | Scale (MAPS20; Côté, 2016) | |
| <b>Exploratory Outcomes</b> | | |
| Subgroup Differences | Baseline Demographic | T1 |
| | Questionnaire | |
| | Session attendance | T1/T2 |
| | Focus group | T2 |
| *Pre-program = T0; Week One = T1; Week Four = T2 | | |

The decision to incorporate the leadership program into an adequately powered definitive trial (alongside rent subsidies and coaching) will be based on feasibility and acceptability. We will not incorporate the leadership program into our planned national larger study if we find program attendance is less than 50%, more than 30% of participants drop out, and/or qualitative feedback from program participants is overwhelmingly negative.

# 2.5 Participant Timeline

We anticipate recruiting participants from June  $3^{rd} - 21^{st}$ , 2024, with a planned program start date of June  $24^{th}$ , 2024 (see Table 3). There will be two sessions/week for four weeks, with a one-week break at the end of Week Two (see Table 1).

Table 3. Schedule of Enrolment, Intervention, and Assessments

| STUDY PERIOD | | | | | |
|---|---|---|---|---|---|
| | Enrolment | Post-enrolment | | | |
| TIMEPOINT | Т0 | T1 | T2 | T3 | T4 |
| | | (Week 1) | (Week 2) | (Week 3) | (Week 4) |
| ENROLMENT: | | L | | | . <b>L</b> |
| Eligibility screening | X | | | | |
| Informed consent | | X | | | |
| INTERVENTION: | | | | | |
| Leadership program | | - | | | <b>—</b> |
| ASSESSMENTS: | | L | | | . <b>L</b> |
| Baseline demographic | | X | | | |
| questionnaire | | | | | |
| Knowledge of program | | X | | | X |
| material | | | | | |
| Identity capital | | X | | | |
| Focus group | | | | | X |
| Program feedback | | | | | X |
| questionnaire | | | | | |

# 2.6 Sample Size

This pilot feasibility and acceptability study was designed with the intention of generating data and hypotheses to inform a national scale-up alongside rent subsidies and coaching. The sample size was pragmatic, based on manageable class sizes and financial resources. No formal sample size calculation was performed.

We plan to enroll 30 youth: 15 from Toronto and 15 from St. Catharines. In addition to purposively recruiting youth (16 - 24 years of age) who have experienced homelessness within the past 12 months, we will target youth who are younger (16 - 18 years of age), identify as girls/women, have a history of being in foster care, and identify as 2SLGBTQ+ given the additional challenges faced by this demographic (see 1. Background and Rationale).

#### 2.7. Recruitment

Study participants will be collaboratively recruited with our long-standing community partners: RAFT (St. Catharines); Covenant House (Toronto); StepStones for Youth (Toronto). RAFT and Covenant House work with young people who are experiencing or have experienced homelessness, and StepStones for Youth works with young people who are in or transitioning out of foster care. Youth will be invited to attend one of two four-week leadership programs – one in St. Catharines and one in Toronto.

Initial introduction to the study will be facilitated by our community partners, and interested participants directed to call or email the study research coordinator (Appendix C: Email and Phone Script). Community partners will utilize the study poster (Appendix D: Study Poster) and consent form (Appendix E: Consent Form) to help guide their initial discussions with potential participants. Screening for eligibility (Table 4) will be done over the phone or via a Zoom call by the research coordinator (Appendix F: Eligibility Screening Script). The eligibility screening checklist will be used verbally for all interested individuals. Notes will only be taken for the purpose of collecting broad, anonymous information about why a potential participant could not meet the eligibility criteria of being able to consistently attend the four-week leadership program, in order to inform our scale-up study (Appendix G: Screening Log). Our team will also record the number of young people deemed ineligible for the study.

**Table 4. Eligibility Screening** 

| | Yes | No |
|---|---|---|
| 16 – 24 years of age (at baseline) | | |
| Have experienced homelessness (e.g., unstable housing arrangements including | | |
| shelter stays, couch surfing, and foster care) for 3 consecutive months in the | | |
| past 12 months | | |
| Able to provide free and informed consent | | |
| Able to speak and read English well enough to give consent and participate in | | |
| the intervention and data collection | | |
| Left homelessness within the past 12 months | | |
| Be able to participate in the four-week, in-person leadership program (attend at | | |
| least 6/8 sessions) | | |
| NOT enrolled in a program or study with similar features to TYOH 2.5 | | |
| MUST SAY "YES" TO ALL TO BE ELIGIBLE FOR ENROLLMENT | | ı |

After eligibility screening, participants will be informed immediately over the phone whether they are eligible or ineligible for the study. If there is any confusion regarding eligibility and/or capacity to consent, the team member will reach out to Dr. Thulien for guidance. In addition to being the study principal investigator, Dr. Thulien is a nurse practitioner with over a decade of experience working exclusively with young people who are experiencing or have experienced homelessness.

Eligible participants will be provided the date/time/location of the first leadership program session. At the beginning of the first session, a research team member will carefully review the consent form with the participants to ensure they have a solid understanding of the study, with particular attention to: 1) overall study aim; 2) study length; 3) data collection; 4) data security; and 5) dissemination. A concerted effort has been made to ensure the consent form is in plain language. Highlighted throughout the document is the fact that informed consent is an ongoing process and can be negotiated at any time.

#### 2.8. Data Collection

To answer *Objective Three* (intervention feasibility and acceptability), we will utilize quantitative measures consisting of recruitment/enrolment/attendance/dropout metrics (see Appendix H: Attendance Log) and a composite program feedback questionnaire along with qualitative measures consisting of focus groups (Tables 2 & 5). To answer *Objective Four* (assessing whether self-reported measures of identity capital and knowledge of program material show improvement immediately post-program compared to baseline), we will utilize MAPS20 (assessment of identity capital; Côté, 2016) and a composite knowledge assessment scale (Tables 2 & 5). To answer *Objective Five* (exploring whether there are differences in outcomes by subgroup and/or program participation levels), we will examine select variables from the baseline demographic questionnaire and attendance/dropout metrics (Tables 2 & 5). Given the differences in time commitment at each data collection session, youth will be paid a data collection honorarium of \$25 at pre-program data collection and \$50 at post-program data collection (Appendix I: Study Budget and Justification).

**Table 5. Quantitative Instruments** 

| Instrument | Psychometric Properties |
|---|---|
| Baseline Demographic Questionnaire | This 18-item self-report measure was |
| | developed for this study and explores |
| | domains related to: age; gender; |
| | race/ethnicity; sexual orientation; immigration |
| | status; child welfare involvement; |
| | homelessness entrenchment; education; social |
| | support; financial support; food security. |
| MAPS20 (Côté, 2016) | This 20-item validated self-report measure |
| | explores domains related to identity capital: |
| | self-esteem; purpose in life; internal locus of |
| | control; self-efficacy/ego strength. Score |
| | range: 20-120; score of less than 71 indicates |
| | risk/vulnerability of being overwhelmed by |
| | any adverse circumstances (internal |
| | consistency of four sub-scales $\alpha = .6175$ ). |
| Knowledge Assessment | This 16-item self-report measure was |
| | developed for this study and explores |
| | domains related to self-leadership such as: |
| | mindfulness; core values; purpose; goal |
| | setting; growth mindset; identity; courage. |
| Composite Program Feedback Questionnaire | This 4-item anonymous questionnaire will be |
| | used to collect information about participants' |
| | view of the leadership program, the impact of |
| | the program on them, and their view of the |
| | individuals running the program. |

# 2.8.1. Quantitative Methods

Quantitative data collection (Appendix J: Quantitative Data Collection Instruments) will be conducted at the beginning of the first leadership program session as well as the last (Tables 3 &

5). T1 (Week One) data collection will consist of: baseline demographic questionnaire; MAPS20 (Côté, 2016); and knowledge assessment. T2 (Week Four) data collection will consist of: MAPS20; knowledge assessment; and program feedback questionnaire. All questionnaires will be completed in-person and on paper.

## 2.8.2. Quantitative Analysis

Quantitative analysis will be conducted using descriptive statistics to measure feasibility and acceptability overall (Objective 3) and by select sub-groups (Objective 5). Non-parametric or t-tests and Cohen's d effect size will be used to examine pre/post leadership program differences in identity capital (MAPS20) and acquired knowledge (Objective 4), and by select sub-groups and program attendance (Objective 5). Biostatistician Dr. Rosane Nisenbaum (co-investigator) will provide oversight to the quantitative data analysis.

## 2.8.3. Qualitative Methods

Qualitative data generation (Appendix K: Focus Group Guide) will take place at the end of the last leadership program session. Each focus group (one in Toronto and one in St. Catharines) will be co-led by Mardi Daley (research team member with lived expertise of homelessness) and Dr. Naomi Thulien and primarily centre around leadership program acceptability (Objective 3). The audio-taped focus groups will last approximately 45-60 minutes. As we have done in previous studies, we will share a nutritious meal together before the focus groups begin, which typically lasts 30-45 minutes. We anticipate 15 young people in each group, divided by location (one group with Toronto youth and one group with St. Catharines youth).

Focus group questions will primarily centre around intervention acceptability but will also explore the impact of the intervention on identity capital (e.g., sense of purpose and control) and socioeconomic inclusion (e.g., connection to broader social networks). The focus groups will be audio recorded using the password-protected application Voice Record Pro on a password-protected device. Audio recordings will be transcribed verbatim by a member of the research team, and the transcripts uploaded to the web-based application Dedoose (SocioCultural Research Consultants, LLC, 2024) for storage and retrieval. One member of the research team will serve as an observer/ note taker at each focus group session to document non-verbal

communication (e.g., eagerness or disinterest) as well as preliminary analytic insights based on listening to the discussion. In addition, each focus group facilitator will document field notes as soon as possible after the meeting to capture their own observations and reflections on the sessions (Luciani et al., 2019; Merriam & Tisdell, 2016).

## 2.8.4. Qualitative Analysis

Qualitative data analysis will be led by Mardi Daley and Dr. Naomi Thulien and conducted using reflexive thematic analysis (Braun & Clarke, 2021) with a critical social theoretical lens (Kirkham & Anderson, 2010; Moosa-Mitha, 2015; Strega, 2015). Briefly, reflexive thematic analysis is part of an analytic process comprised of six iterative phases (data familiarization, coding, initial theme generation, theme development and review, theme refining, and writing up) that also requires engagement with theory, reflexivity (acknowledging the role of the researcher in shaping the findings), and interpretation (i.e., not expecting the data to 'speak for itself') (Luchenski et al., 2018). A critical social theoretical lens will help the team use an intersectional approach to uncover and speak about inequitable societal factors that may disproportionately impact some youth (e.g., youth who identify as 2SLGBTQ+ or girls/women) while also highlighting participants' individual strengths despite these inequities (Kirkham & Anderson, 2010; Moosa-Mitha, 2015; Strega, 2015).

Prior to the first qualitative data analysis session, two team members will read the two focus group transcripts multiple times, code data relevant to intervention acceptability and our assumption that identity capital is a mitigating factor in socioeconomic inclusion (and look for data that might disprove this assumption), and compare codes across both transcripts (Bhattacharya, 2017; Creswell & Creswell, 2017; Luciani et al., 2019). During the analysis sessions, the codes will be discussed (and revised/deleted as needed) and organized in a code book, clustered into categories, and eventually synthesized into key themes. Analysis will primarily be inductive (moving from data to conceptualizing); however, deductive reasoning (moving from conceptualizing to data) will be employed when we want to understand new data through the lens of our emerging conceptual framework. Preliminary data analysis will be discussed with youth advisors and their feedback will be incorporated into further analysis and

interpretation, collaborative knowledge mobilization, and co-planning a national scale-up (alongside rent subsidies and coaching).

## 2.9. Data Monitoring

As is common in pilot and feasibility studies, there is no interim quantitative analysis planned to guide a decision to stop the study early (Eldridge et al., 2016). That said, at least one member of our research team will attend every leadership session to monitor participant engagement. We will consider making adjustments to the leadership program if informal feedback from participants is overwhelmingly negative and/or the majority of young people stop participating.

## 3. Limitations

This study has limitations. First, this is a feasibility and acceptability study and thus not adequately powered to detect a significant difference in quantitative self-report measures; results must be interpreted with caution. Second, all young people will be connected to urban-based social service agencies in the province of Ontario; youth living in rural locations and/or outside of Ontario may not take up the program in the same way. Third, all of the quantitative instruments are based on self-reports and thus subject to social desirability bias. Finally, the quantitative measures we have developed/chosen are what we believe will capture knowledge of self-leadership and identity capital; it is plausible that these measures do not adequately capture these domains with this population.

## 4. Ethics and Dissemination

We have endeavoured to weave ethical considerations into all aspects of the study design, including our decision to utilize a CBPAR methodology, which foregrounds community (especially youth) priorities. The decision to conduct this leadership program was a direct result of feedback from youth in our current TYOH 2.0 study. In addition, we have fostered relationships with our youth advisors over the past five years, and they were actively involved in developing this protocol. Ethical approval for this study will be obtained by the Unity Health Toronto Research Ethics Board.

## 4.1. Risks, Benefits, and Safety

Given the nature of this strengths-based leadership program and our close relationship with the TYOH 2.5 program coaches (also coaches in our TYOH 2.0 study), we believe the harms and risks to participants will be minimal. While we have intentionally not chosen deficit-focused questions/scales for the quantitative questionnaires, it is plausible that some participants could find certain questions distressing. For this reason, participants will be informed that they can skip questions if they choose, or stop the questionnaire at any time. The focus group questions will also target participant strengths; however, participants will be reminded at the start of each session that they do not have to answer any questions that make them uncomfortable. They will also be reminded that we cannot guarantee other focus group members will not share discussion topics outside of the focus group sessions. As noted in the consent form, participants will be made aware that they may withdraw from the study at any time.

Coaches and participants will also be provided with a mental health resource document (see Appendix L: Mental Health Resources) to utilize as needed. The study team/coaches will reach out to Dr. Thulien to discuss a case if there are any concerns related to mental health distress. Dr. Thulien will reach out to community partners at RAFT (St. Catharines), StepStones for Youth (Toronto), and/or Covenant House Toronto to help connect youth to psychosocial supports as needed. We have employed a similar strategy with our community partners for the past seven years. In our experience, these cases are rare, and our management plan has worked well.

All participants will likely benefit from participating in the weekly leadership sessions.

Participants may also benefit from having the opportunity to contribute their expertise during the focus group sessions; this has been our experience with previous studies.

## 4.2. Confidentiality

Privacy and confidentiality considerations have been woven throughout the research process:

- 1. <u>Recruitment:</u> Interested participants will reach out to the lead research coordinator directly rather than community partners sharing contact information with the team.
- 2. <u>Eligibility screening:</u> No personal health information or personal identifying information will be collected.

- 3. <u>Enrollment:</u> Consent will be required prior to baseline data collection. The consent form indicates that limits to confidentiality apply if a participant discloses that they intend to hurt themselves or others, or if they inform a member of the research team that someone under the age of 16 years is suffering abuse and/or neglect.
- 4. <u>Quantitative data collection:</u> Paper copies of the consent forms and questionnaires will be stored in a locked filing cabinet at the MAP Centre for Urban Health Solutions in an area only accessible to those with electronic and key access.
- 5. Qualitative data collection: Focus groups will be audio recorded on a password-protected application and on a password-protected device. The audio-recorded files will be securely sent to a research team member via Unity Health email with a link that expires in 24 hours. After the team member has transcribed the audio file, they will delete the file. All transcripts will be stored on a SMH secure server and uploaded to Dedoose (SocioCultural Research Consultants, LLC, 2024). Pseudonyms will be used in place of real names in focus group transcripts.
- 6. <u>Linking log:</u> A key that links each participant's name with their participant identification number will be created by the lead research coordinator and stored as a separate electronic file on the SMH secure serve (Appendix M: Linking Log).
- 7. <u>Data access:</u> Only authorized members of the research team will have access to quantitative and qualitative study data, and an access log will be maintained by the lead research coordinator. De-identified raw data will be made available upon reasonable request (e.g., request comes from a researcher affiliated with an academic institution).
- 8. <u>Data retention:</u> All data will be destroyed after 7 years. Dr. Thulien will be responsible for ensuring the data is destroyed.

#### 4.3. Dissemination

Our team is committed to diverse and accessible forms of knowledge mobilization. For example, Dr. Thulien was the executive director on the documentary film Searching for Home, which followed three participants from TYOH 1.0 (<a href="www.searchingforhome.ca">www.searchingforhome.ca</a>). Dr. Thulien also coproduced a five-minute animation (<a href="www.searchingforhome.ca">www.searchingforhome.ca</a>) about TYOH 1.0 findings. Key mobilization activities for this project include collaborating with youth advisors on dissemination

to multisectoral stakeholders through plain language reports, policy briefs, social media, op-eds, academic and non-academic presentations, and at least one publication in an open-access journal.

# 4.4. Significance

If this leadership program shows promise, we plan to take findings from this project and: 1) incorporate them into a national scale-up alongside rent subsidies and coaching; 2) explore offering the leadership program in settings such as schools and/or community-based after-school programs; 3) co-share broadly with frontline workers, educators, and policymakers the value in targeting the inequitable distribution of identity capital as part of a homelessness prevention strategy.

#### References

Abramovich, A. (2016). Preventing, reducing and ending LGBTQ2S youth homelessness: The need for targeted strategies. *Social Inclusion*, 4(4), 86–96. <a href="https://doi.org/10.17645/si.v4i4.669">https://doi.org/10.17645/si.v4i4.669</a>

Bhattacharya, K. (2017). Fundamentals of qualitative research: A practical guide. Routledge.

Bonakdar, A., Gaetz, S., Banchani, E., Schwan, K., Kidd, S., O'Grady, B. (2023). Child protection services and youth experiencing homelessness: Findings of the 2019 national youth homelessness survey in Canada. *Children and Youth Services Review*, *153*(107088), 1–8. <a href="https://doi.org/10.1016/j.childyouth.2023.107088">https://doi.org/10.1016/j.childyouth.2023.107088</a>

Braun, V., & Clarke, V. (2021). Thematic analysis: A practical guide. SAGE.

Brueckner, M., Green, M., & Saggers, S. (2011). The trappings of home: Young homeless people's transitions towards independent living. *Housing Studies*, *26*(1), 1–16. https://doi.org/10.1080/02673037.2010.512751

Centrepoint. (2022). Policy and research: Our research. <a href="https://centrepoint.org.uk/research-reports">https://centrepoint.org.uk/research-reports</a>

ClinicalTrials.gov. (2023). Transitioning youth out of homelessness 2.0 (TYOH 2.0). <a href="https://clinicaltrials.gov/study/NCT05781503">https://clinicaltrials.gov/study/NCT05781503</a>

Côté, J. (2016). *The identity capital model: A handbook of theory, methods, and findings*. https://ir.lib.uwo.ca/cgi/viewcontent.cgi?article=1038&context=sociologypub.

Crandall, A., Miller, J. R., Cheung, A., Novilla, L. K., Glade, R., Novilla, M. L. B., Magnusson, B. M., Leavitt, B. L., Barnes, M. D., & Hanson, C. L. (2019). ACEs and counter-ACEs: How positive and negative childhood experiences influence adult health. *Child Abuse & Neglect*, *96*(104089), 1–9. <a href="https://doi.org/10.1016/j.chiabu.2019.104089">https://doi.org/10.1016/j.chiabu.2019.104089</a>

Creswell, J. W., & Creswell, J. D. (2017). Research design: Qualitative, quantitative, and mixed methods approaches. SAGE.

Dej, E. (2020). A complex exile: Homelessness and social exclusion in Canada. UBC Press.

Eldridge, S. M., Chan, C. L., Campbell, M. J., Bond, C. M., Hopewell, S., Thabane, L., Lancaster, G. A., & PAFS consensus group (2016). CONSORT 2010 statement: Extension to randomised pilot and feasibility trials. *BMJ*, *355*(i5239), 1–29. https://doi.org/10.1136/bmj.i5239

Gaetz S, O'Grady B, Kidd S, Schwan K. (2016). Without a home: The national youth homelessness survey. Canadian Observatory on Homelessness Press. https://homelesshub.ca/sites/default/files/WithoutAHome-final.pdf

Israel, B. A., Schulz, A. J., Parker, E. A., Becker, A. B., Allen, A. J., Guzman, J. R., & Lichtenstein, R. (2018). Critical issues in developing and following CBPR principles. In N. Wallerstein, B. Duran, J. Oetzel, & M. Minkler (Eds.). *Community-based participatory research for health: Advancing social and health equity* (3<sup>rd</sup> ed., pp. 31–46). Jossey-Bass.

Karabanow, J. (2004). Being young and homeless: Understanding how youth enter and exit street life. Peter Lang Publishing.

Karabanow, J., Kidd, S., Frederick, T., & Hughes, J. (2016). Toward housing stability: Exiting homelessness as an emerging adult. *The Journal of Sociology & Social Welfare, 43*(1), 121–148. https://doi.org/10.15453/0191-5096.4000

Kidd, S. A., Frederick, T., Karabanow, J., Hughes, J., Naylor, T., & Barbic, S. (2016). A mixed methods study of recently homeless youth efforts to sustain housing and stability. *Child and Adolescent Social Work Journal*, *33*(3), 207–218. <a href="https://doi.org/10.1007/s10560-015-0424-2">https://doi.org/10.1007/s10560-015-0424-2</a>

Kidd, S. A., Gaetz, S., O'Grady, B., Schwan, K., Zhao, H., Lopes, K., & Wang, W. (2021). The second national Canadian homeless youth survey: Mental health and addiction findings. *Canadian Journal of Psychiatry*, 66(10), 897–905. <a href="https://doi.org/10.1177/0706743721990310">https://doi.org/10.1177/0706743721990310</a>

Kirkham, S. R., & Anderson, J. M. (2010). The advocate-analyst dialectic in critical and postcolonial feminist research: Reconciling tensions around scientific integrity. *Advances in Nursing Science*, *33*(3), 196–205. https://doi.org/10.1097/ANS.0b013e3181e4a7d3

Kozloff, N., Adair, C. E., Palma Lazgare, L. I., Poremski, D., Cheung, A. H., Sandu, R., & Stergiopoulos, V. (2016). "Housing First" for homeless youth with mental illness. *Pediatrics*, *138*(4), 1–10. <a href="https://doi.org/10.1542/peds.2016-1514">https://doi.org/10.1542/peds.2016-1514</a>

Liu, M., Luong, L., Lachaud, J., Edalati, H., Reeves, A., & Hwang, S. W. (2021). Adverse childhood experiences and related outcomes among adults experiencing homelessness: A systematic review and meta-analysis. *Lancet Public Health*, *6*(11), e836–e847. <a href="https://doi.org/10.1016/S2468-2667(21)00189-4">https://doi.org/10.1016/S2468-2667(21)00189-4</a>

Luchenski, S., Maguire, N., Aldridge, R. W., Hayward, A., Story, A., Perri, P., Withers, J., Clint, S., Fitzpatrick, S., & Hewett, N. (2018). What works in inclusion health: overview of effective interventions for marginalised and excluded populations. *Lancet*, *391*(10117), 266–280. https://doi.org/10.1016/S0140-6736(17)31959-1

Luciani, M., Campbell, K., Orr, E., Nguyen, L., Manja, V., Ausili, D., & Jack, S. M. (2019). How to design a qualitative health research study. Part 2: Data generation and analysis considerations. *Professioni Infermieristiche*, 72(3), 221–231.

Mayock, P., O'Sullivan, E., Corr, M.L. (2011). Young people exiting homelessness: An exploration of process, meaning and definition. *Housing Studies*, *26*(6), 803–826. https://doi.org/10.1080/02673037.2011.593131

Merriam, S. B., & Tisdell, E. J. (2015). *Qualitative research: A guide to design and implementation*. John Wiley & Sons.

Moosa-Mitha, M. (2015). Situating anti-oppressive theories within critical and difference-centred perspectives. In S. Strega & L. Brown (Eds.). *Research as resistance: Critical, Indigenous, & anti-oppressive approaches* (2<sup>nd</sup> ed., pp. 65–95). Canadian Scholars Press.

Morton, M. H., Dworsky, A., Matjasko, J. L., Curry, S. R., Schlueter, D., Chávez, R., & Farrell, A. F. (2018). Prevalence and Correlates of Youth Homelessness in the United States. *The Journal of Adolescent Health*, *62*(1), 14–21. https://doi.org/10.1016/j.jadohealth.2017.10.006

Morton, M. H., Kugley, S., Epstein, R., & Farrell, A. (2020). Interventions for youth homelessness: A systematic review of effectiveness studies. *Children and Youth Services Review*, *116*(105096), 1–13. <a href="https://doi.org/10.1016/j.childyouth.2020.105096">https://doi.org/10.1016/j.childyouth.2020.105096</a>

Samuels, G.M., Cerven, C., Curry, S., Robinson, SR., Patel, S. (2019). Missed opportunities in youth pathways through homelessness. <a href="https://www.chapinhall.org/wp-content/uploads/ChapinHall\_VoYC\_Youth-Pathways-FINAL.pdf">https://www.chapinhall.org/wp-content/uploads/ChapinHall\_VoYC\_Youth-Pathways-FINAL.pdf</a>

SocioCultural Research Consultants, LLC. (2024). Dedoose Version 9.2.006, web application for managing, analyzing, and presenting qualitative and mixed method research data. https://www.dedoose.com/

Strega, S. (2015). The view from the Poststructural margins: Epistemology and methodology reconsidered. In S. Strega & L. Brown (Eds.). *Research as resistance: Critical, Indigenous, & anti-oppressive approaches* (2<sup>nd</sup> ed., pp. 119-152). Canadian Scholars Press.

Thulien, N. S., Amiri, A., Hwang, S. W., Kozloff, N., Wang, A., Akdikmen, A., Roglich, J., & Nisenbaum, R. (2022). Effect of portable rent subsidies and mentorship on socioeconomic inclusion for young people exiting homelessness: A community-based pilot randomized clinical trial. *JAMA Network Open*, 5(10), 1–13. https://doi.org/10.1001/jamanetworkopen.2022.38670

Thulien, N. S., Gastaldo, D., Hwang, S. W., & McCay, E. (2018). The elusive goal of social integration: A critical examination of the socio-economic and psychosocial consequences experienced by homeless young people who obtain housing. *Canadian Journal of Public Health*, 109(1), 89–98. https://doi.org/10.17269/s41997-018-0029-6

Thulien, N. S., Hwang, S. W., Kozloff, N., Nisenbaum, R., Akdikmen, A., Fambegbe, O. P., Feraday, R., Mathewson, C., Mutamiri, M., Roglich, J., Wang, A., Zagala, M., & Amiri, A. (2023). "When I think about my future, I just see darkness": How youth exiting homelessness navigate the hazy, liminal space between socioeconomic exclusion and inclusion. *Canadian Journal of Public Health*, *114*(6), 893–905. <a href="https://doi.org/10.17269/s41997-023-00804-2">https://doi.org/10.17269/s41997-023-00804-2</a>

Thulien, N. S., Kozloff, N., McCay, E., Nisenbaum, R., Wang, A., & Hwang, S. W. (2019). Evaluating the effects of a rent subsidy and mentoring intervention for Youth Transitioning Out of Homelessness: Protocol for a mixed methods, community-based pilot randomized controlled trial. *JMIR Research Protocols*, 8(12), 1–11. <a href="https://doi.org/10.2196/15557">https://doi.org/10.2196/15557</a>